CLINICAL TRIAL: NCT02199262
Title: Quality Improving Program on Agitation in the Surgical Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Pr. Bara RICOU, Professor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CER:02-190
Record Dates: First submitted 2014-07-17; First posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Agitation
Keywords: Intensive care unit; Incidents; prevention; music; reflexology
MeSH Terms: conditions — Psychomotor Agitation | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- control groupe (Experimental): agitation diagnosis and management according to implemented guidelines= reminder implementation
  Interventions: Other: reminder
- music intervention + reminder (Experimental): agitation diagnosis and management according to implemented guidelines+ music intervention
  Interventions: Other: music intervention
- reflexology + reminder (Experimental): agitation diagnosis and management according to implemented guidelines + reflexology
  Interventions: Other: reflexology

INTERVENTIONS:
Other: music intervention — reminder+ 20 minutes in the morning and 20 minutes in the afternoon of music listening(classical or soft background music), delivered by compact disc players with headphones with disposable ear pads.
  Arms: music intervention + reminder
Other: reflexology — reminder + 20 minutes per day feet reflexology massage provided by certified specialist in reflexology massages
  Arms: reflexology + reminder
Other: reminder — Implementation of a reminder of guidelines of agitation diagnosis and management
  Arms: control groupe

SUMMARY:
Agitation in the intensive care unit can have multiple consequences. The investigators hypothesize that agitation and its consequences can be reduced by the introduction of a reminder aiming at guiding the management of agitation. The investigators also hypothesize that they can prevent agitation and its consequences by acting on patients environment with reafferentation and relaxation methods.

The investigators' objectives are to test within a quality improvement project by a prospective randomized study:

* If by reducing the number of agitation episodes we reduce the number of harmful consequences.
* If the introduction of reafferentation and relaxation methods (music therapy or reflexology) can prevent the occurrence of agitation.
* If the introduction of a reminder on management of agitation can reduce the number of agitation episodes.

This study is conducted in an18 general surgical ICU beds receiving 1600 patients / year for a total of 6900 hospital /days /year, in a tertiary teaching hospital.

The study is organized in 3 phases:

1. First phase: Baseline phase (Prospective analysis of the present situation)
2. Second phase: Learning phase (Implementation of a reminder about the management of agitation and delirium )
3. Third phase: Randomized Intervention (reminder alone vs addition of music or reflexology)

The interventions are :

1. Implementation of a reminder of guidelines of agitation diagnosis and management.
2. Music intervention( see description below) + reminder
3. Reflexology (see description below)+ reminder

Agitation is monitored with two scales SAS and CAM-ICU(description below) . Harmful consequences and complications are systematically registered as well as medication and the use of contention methods.

Adherence to the implemented monitoring and interventions is also regularly checked.

Data are daily collected (see details below) Statistical analysis and power calculation (see below)

DETAILED DESCRIPTION:
Agitation in the intensive care unit (ICU) can be described as an excessive, usually no purposeful motor activity associated with internal tension.Agitation can have multiple consequences.

The occurrence of agitation episodes is a problem recognized for several years and already widely discussed in the literature.

Delirium is a reversible, global impairment of cognitive processes, usually of sudden onset, coupled with disorientation, impaired short term memory, altered sensory perception (hallucinations), abnormal thought process, and inappropriate behavior.

The analysis of the literature and a previous pilot study in the unit brought us to the consideration that a quality assessment and improvement project should be started aiming at monitoring and influencing the occurrence of agitation and their consequences such as the morbidity and mortality of the patients, the impact on care delivery and maybe the economic repercussions.

Investigators hypothesized that agitation and its consequences can be reduced by the introduction of a reminder aiming at guiding the management of agitation. While the optimization of the management of the related states (such as delirium, pain and anxiety) is crucial, investigators hypothesized that we could prevent agitation and its consequences by acting on patients environment with reafferentation and relaxation methods.

The investigators' objectives will be to test within a quality improvement project by a prospective randomized study:

* If by reducing the number of agitation episodes we reduce the number of harmful consequences.
* If the introduction of reafferentation and relaxation methods (music therapy or reflexology) can prevent the occurrence of agitation.
* If the introduction of a reminder on management of agitation can reduce the number of agitation episodes.

Setting:

18 general surgical ICU beds receiving 1600 patients / year for a total of 6900 hospital /days /year, in a tertiary teaching hospital. The ICU is divided in 6 rooms with 3 beds: 1 at the window, 1 in the middle of the room and 1 by the room door. Each room has one clock in front of the central bed.

The nurse to patient ratio is during daytime 1:1.5 and 1:2 during nighttime. Nurses working shifts are organized in 3 times 8 hours every day. This study has been approved by the head of division and will be conducted solely inside the surgical ICU. As a quality improvement program, no consent by patients is required, according to the CEREH /HUG recommendations.

Patients:

Investigators will enroll every patient older than 18 years staying more than 24 hours in the ICU

1. First phase: Baseline phase (Prospective analysis of the present situation)
2. Second phase: learning phase (Implementation of a reminder about the management of agitation and delirium )
3. Third phase: Randomized Intervention (reminder alone vs addition of music or reflexology)

Interventions:

Reminder :

The care giver will be helped in the diagnosis of the cause, the management of and the treatment of agitation and delirium by a reminder. This reminder has been adapted from the guidelines from the ACCP and SCCM comity. It has been adapted on local needs by a multidisciplinary group including nurses and physicians from the ICU. Investigators will instruct nurses and physicians on the use of the reminder 3 times a week for 20 min during 1 month. Investigators will provide pocket reminders for every care giver and display posters of the reminder in key points of the ICU. The reminder will also be available on the intranet site and introduced in the SISIF system (bedside computerized patient chart).

The music intervention consisted in two daily sessions of at least 20 minutes music listening ( classical and soft background music ) .The music intervention was delivered by compact disc players with headphones with disposable ear pads.

The reflexology is a feet massage technique consisting in massages and pressures on precise points of the feet.This therapy was applied for 20 minutes each day to the ICU patients by a certified specialist in reflexology massage

Indicators :

Indicators of agitation:

1.Sedation Agitation scale (SAS) and Confusion Assessment Method for ICU (CAM-ICU): The SAS scale is recognized for its reliability and validity for the sedation and agitation assessment. It is a single item scale graded from 1 (coma) to 7 (extremely agitated. Agitation is diagnosed if SAS >4.

The CAM-ICU score is a modified version of the CAM scale adapted to intensive care patients. This scale assesses delirium (positive CAM-ICU test) by considering four different parameters that mostly focus on patient's cognitive state . It is also validated and recognized for its high specificity and sensitivity.

Investigators will analyze the presence or absence of delirium at each evaluation judged necessary by the nurse, at least once by shift (every 8 hours).

Investigators will then investigate whether 1. the positive CAM-ICU will precede the occurrence of agitation defined as SAS>4, 2. whether low values of SAS, <4 or >4 precede higher values of SAS.

Indicators of the harmful consequences:

1. Complications : Investigators will register the events related to an agitation episode or delirium and classify them in three groups. The three groups are determined by the potential life threatening character of the event. One event can be considered as severe i.e. really life threatening (self extubation, ventilator disconnection, central catheter removal, chest tube removal, trauma, falling from bed), moderate (removal of nasogastric tube, peripheral venous or arterial catheter) or mild i.e. not life threatening (contortion of the patient in his bed, patient's aggressiveness toward the staff, urethral catheter removal, electrode or saturation monitoring removal).
2. Medication : Investigators will register the patient's medication in a daily total dose (mg /patient/day/drug) of 3 drug groups in relation with agitation. Investigators will compare the use of medication during the different study phases and between the 3 different groups during the third phase.

   sedatives: oxazepam, lorazepam,midazolam, propofol analgesics: acetaminophen, ibuprofen, morphine, fentanyl, ketorolac antipsychotics: haloperidol, thioridazine
3. The use of contention methods will be registered will be compared for each phase of the study.

Indicators of adherence:

1. Adherence to the implementation of monitoring (SAS, CAM-ICU) during the 3 phases.
2. Adherence to the reminder
3. Adherence to intervention (reflexology and music therapy)

Indicators of safety:

Investigators will assess the occurrence of adverse events potentially related to the therapy or management of agitation.

1. Intubations: the study team will register the number of intubations related to agitation.
2. Antagonist drugs: the study team will register the use of antagonist drugs such as naloxone chlorhydrate (Narcan®), flumazenil (Anexate®) and biperidene(Akineton®) following the treatment of agitation .

Data collection First phase

1. 24 hours after ICU admission, the study team will assess the demographic and actual diagnostic data, the past medical history, the usual and actual treatment, the current smoking history, alcohol and drug abuse, the invasive equipment and the APACHE II score.
2. Daily investigators will also assess the treatment and equipment modifications, the laboratory values of variables potentially related to agitation (sodium, glucose, calcium, urea, creatinine, bilirubin, oxygen saturation, FiO2), fever, the occurrence of infections, the introduction of therapeutic antibiotics. The bed location in the room will be specified (door, middle, window). Investigators will also daily record the consequence (annex 7) and safety indicators . No additional test or exam will be performed for the purpose of the study.
3. Three times a day (once by nurse shift) the nurses will assess agitation and delirium by SAS and CAM-ICU. Each time the attending nurse notices a modification of degree of agitation, she will register the concomitant SAS.
4. At the end of each patient stay investigators will calculate the total dosage (mg/kg/day) p.o. or i.v of sedatives (benzodiazepines, propofol or others), analgesics (acetaminophen, NSARs, morphine, fentanyl or others) or antipsychotic drugs (haloperidol or others) delivered to every patient.

Second phase In addition to all the data collected during the first phase, investigators will register the adherence to the reminder at each agitation episode.

Third phase Same data as during the second phase. In addition, investigators will note daily the correct delivery of the allocated intervention.

Statistical analysis and power calculation:

Investigators will use analysis of variance (ANOVA) with Bonferroni's post-test or Kruskal-Wallis where appropriated. Proportions will be analyzed by Pearson's 2.

The endpoint of the study is to reduce the occurrence of the consequences of agitation and/or delirium. The sample size is calculated to detect a minimum mean difference of 50% of the number of patient days with occurrence of the consequences of agitation and delirium. In a preliminary study, investigators assessed the occurrence of "consequences" in about 20% of patient/days.

The number (=n) of patients needed to detect a minimum mean difference of 50% between the baseline and the learning phase is 219 (a 0.05, power 80% two sided), and 219 in the three randomization groups. 80 patients per month present the inclusion criteria for the study. Thus, we need 2.7 months in the Baseline, a minimum of 2.7 months in the Learning and 8.1 months for the Randomization Intervention periods.

All continuous variables will be expressed as mean SD (normally distributed) or medians and range (non normally distributed). A p value <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* admission in ICU >24 hours

Exclusion Criteria:

* amputation
* paraplegia
* non french speaking
* consent refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1107 (Actual)
Dates: Start 2004-02; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Diminution of agitation (SAS and CAM-ICU) trough a music intervention or reflexology | lenght of patients' stay, 3.5 days on average
  Music intervention: The patient will listen to a variety of music for at least 20 minutes in the morning and in the afternoon (compact disc players with headphones with disposable ear pads). The preferred music will be freely available for the rest of the day. The choice of the music type will depend on the patients ability to communicate his desires. If the patient is not able to express his choice, the caregiver will ask his next of kin. If the information is not available, the caregiver will select a type of music he judges adapted to the patient's situation.
  Reflexology: This therapy will be applied 20 minutes per day to patients by a certified specialist in reflexologic massages.
  Measurements : Investigators analyze the presence or absence of agitation and delirium by SAS and CAM-ICU at each evaluation judged necessary by the nurse, at least once by shift (every 8 hours).

SECONDARY OUTCOMES:
Correlation between the reduction of the number of agitation episodes (SAS and CAM-ICU) and the number of harmful consequences | lenght of patients' stay, 3.5 days on average
  1. Complications : Investigators will register the events related to an agitation episode or delirium and classify them in three groups determined by the potential life threatening character of the event. One event can be considered as severe i.e. really life threatening (self extubation, ventilator disconnection, central catheter removal, chest tube removal, trauma, falling from bed), moderate (removal of nasogastric tube, peripheral venous or arterial catheter) or mild i.e. not life threatening (contortion of the patient in his bed, patient's aggressiveness toward the staff, urethral catheter removal, electrode or saturation monitoring removal).
  2. Medication : Investigators will register the patient's medication in a daily total dose (mg /patient/day/drug) of 3 drug groups in relation with agitation (sedatives, analgesics, antipsychotics).
  3. The use of contention methods will be registered will be compared for each phase of the study.

OTHER OUTCOMES:
Effect of reminder of guidelines of agitation diagnosis (by SAS and CAM-ICU ) and management | lenght of patients' stay, 3.5 days on average
  The caregiver will be helped in the diagnosis of the cause, the management of and the treatment of agitation and delirium by a reminder. This reminder has been adapted from the guidelines from the ACCP and SCCM committee. Investigators will instruct nurses and physicians on the use of the reminder 3 times a week for 20 min during 1 month. Investigators will provide pocket reminders for every caregiver and display posters of the reminder in key points. The reminder will also be available on the intranet site and introduced in the SISIF system (bedside computerized patient chart).
  Measurement: At each agitation episode, the physician in charge of the patient will be asked the etiology of the agitation. The treatment chosen according to this diagnosis will be compared to the treatment proposed in the reminder. The percentage of treatment conforming to the reminder will be considered as the adherence to the reminder.

CONTACTS AND LOCATIONS:
Locations (1):
- Surgical Intensive Care Unit, Geneva, Canton of Geneva, Switzerland